CLINICAL TRIAL: NCT04921709
Title: Evaluation of Renal Involvement in Inflammatory Bowel Disease Patients
Brief Title: Renal Involvement in Inflammatory Bowel Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Hamdy Tawfik Abdelhakim, Principal Investigator, Assiut University
Other Study IDs: IBD impacts on kidney
Record Dates: First submitted 2021-03-03; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD Patients with Renal Involvement: 1. Inclusion criteria: - patients with IBD diagnosed by colonoscopy and histopathology will classify the activity of the case to mild ,moderate and severe according to Mayo classification and have renal problems .
     Age (18-65 years)
  2. Exclusion criteria: 1-patients underage of 18 2-HCV or HBV patients 3- renal patients diagnosed before diagnosis of IBD 4- diabetic or hypertensive patients 5- other autoimmune diseases such as Rheumatoid Arthritis, SLE. 6- Malignancy
  Interventions: Other: Medical tests
- IBD Patients without Renal Involvement: 1. Inclusion criteria: - patients with IBD diagnosed by colonoscopy and histopathology will classify the activity of the case to mild ,moderate and severe according to Mayo classification and have no renal problems .
     Age (18-65 years)
  2. Exclusion criteria: 1-patients underage of 18 2-HCV or HBV patients 3- renal patients diagnosed before diagnosis of IBD 4- diabetic or hypertensive patients 5- other autoimmune diseases such as Rheumatoid Arthritis, SLE. 6- Malignancy
  Interventions: Other: Medical tests

INTERVENTIONS:
Other: Medical tests — Blood tests

SUMMARY:
To evaluate renal involvement in inflammatory bowel disease patients .

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic, relapsing and remitting inflammatory condition predominantly affecting the gastrointestinal (GI) tract that results from complex interplay of the individual's genetic makeup, the environment, the gut microbiota and the host immune response .

IBD is an umbrella disorder that covers Crohn's disease, ulcerative colitis and IBD unclassified . Crohn's disease is characterised by transmural inflammation that can affect any part of the GIT with characteristic skip lesions of healthy tissues, while ulcerative colitis is a continuous mucosal inflammation largely confined to the colon. 'IBD unclassified' is a term used when the endoscopic and histological features are not sufficient to favour one of the other diagnoses.

The prevalence of extraintestinal manifestations (EIMs) in inﬂammatory bowel diseases (IBDs) varies from 6%-46%.

The mechanisms that have been suggested include contributions of genetic factors, infectious agents, circulating bacterial endotoxins and immune-complex deposition.

EIMs can involve almost every organ system. It is not always possible to identify the pathophysiological mechanism underlying an organ's involvement in IBD; it may originate from the same pathophysiological mechanism as intestinal disease, or as a secondary complication of IBDs, Renal involvement has been considered as an EIM and has been described both in Crohn's disease (CD) and in ulcerative colitis (UC).

Renal EIMs and IBD-related therapy are potential risk factors for the development of renal insufficiency (both acute and chronic) in patients with CD and UC.

Chronic kidney disease (CKD) is a type of kidney disease in which there is gradual loss of kidney function over a period of months to years.

CKD is defined as kidney damage or glomerular filtration rate (GFR) <60 ml /min/1.73 m2 for 3 months or more .

GFR can be estimated from calibrated serum creatinine and estimating equations ,such as the Modification of Diet in Renal Disease (MDRD) study equation or the Cockcroft -Gault formula .

Kidney disease severity is classified into five stages according to the level of GFR.

1. Stage 1: Slightly diminished function; kidney damage with normal or relatively high GFR (≥90 ml/min/1.73 m2)
2. Stage 2: Mild reduction in GFR (60-89 ml/min/1.73 m2) with kidney damage
3. Stage 3: Moderate reduction in GFR (30-59 ml/min/1.73 m2)
4. Stage 4: Severe reduction in GFR (15-29 ml/min/1.73 m2)
5. Stage 5: Established kidney failure (GFR <15 ml/min/1.73 m2)

The most frequent renal diseases in patients with IBD are: nephrolithiasis, tubulointerstitial nephritis, glomerulonephritis and amyloidosis .

As in other EIMs, renal manifestations can be considered as dependent on the same immunological mechanism that determines intestinal inﬂammatory diseases, directly related to intestinal activity. Another hypothesis to be considered is that renal involvement is an independent of bowel disease, due to its autoimmune mechanism of action; otherwise, it could be related to metabolic disorders that develop in IBD. Finally, kidney pathologies in IBD have been associated with side e!ects of drugs Aminosalicylates, azathioprine, cyclosporin and TNFα inhibitors may be involved in renal impairment. However, it is not always possible to clarify the mechanism of these drugs in kidney damage. In many cases it remains unclear whether renal impairment is an EIM or a drug adverse effect

ELIGIBILITY:
Inclusion Criteria:

* patients with IBD diagnosed by colonoscopy and histopathology will classify the activity of the case to mild ,moderate and severe according to Mayo classification and have renal problems .
* Age (18 - 65 years)

Exclusion Criteria:

* patients underage of 18
* HCV or HBV patients
* renal patients diagnosed before diagnosis of IBD
* diabetic or hypertensive patients
* other autoimmune diseases such as Rheumatoid Arthritis, SLE.
* Malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cohort study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
correlation between lab, radiological and colonoscopy | Baseline
  All patients will be subjected to full clinical history , examination and investigation
  .investigations will include:
  A-Laboratory tests:
  * CBC
  * urine analysis
  * calculating the estimated glomerular filtration rate (eGFR)
  * 24hr urinary protein
  * hepatitis markers ,liver function tests
  * kidney function tests.
  * -kidney biopsy for patients with renal involvement if needed
  * ANA, Anti ds
  * blood electrolyte ( Na, K, Ca , Mg ) B- Radiological: abdominal ultrasonography C- colonoscopy . to evaluate renal ivolvement in inflammatory bowel disease

CONTACTS AND LOCATIONS:
Overall Officials: Enas A Reda Alkaremy, Prof, Study Director — Alkareemy@yahoo.com
Locations (1):
- Hend Hamdy Tawfik, Minya, Egypt

REFERENCES:
- [Background] Oikonomou K, Kapsoritakis A, Eleftheriadis T, Stefanidis I, Potamianos S. Renal manifestations and complications of inflammatory bowel disease. Inflamm Bowel Dis. 2011 Apr;17(4):1034-45. doi: 10.1002/ibd.21468. Epub 2010 Sep 14. PMID 20842645
- [Background] Pardi DS, Tremaine WJ, Sandborn WJ, McCarthy JT. Renal and urologic complications of inflammatory bowel disease. Am J Gastroenterol. 1998 Apr;93(4):504-14. doi: 10.1111/j.1572-0241.1998.156_b.x. PMID 9576439
- [Background] Yoo YJ, Chung SY, Gu DH, Ko GJ, Pyo HJ, Kwon YJ, Bak YT, Won NH. A case of late onset-acute tubulointerstitial nephritis with infliximab and mesalazine treatment in a patient with Crohn's disease. Korean J Gastroenterol. 2014 May;63(5):308-12. doi: 10.4166/kjg.2014.63.5.308. PMID 24870303